CLINICAL TRIAL: NCT02144844
Title: A Behavioral Intervention to Reduce Risk of Antepartum Depression
Brief Title: A Public Health Program to Reduce Risk of Antepartum Depression
Acronym: APD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: East Carolina University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Darlene Elizabeth Jesse, Professor, East Carolina University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 8045091; 1R34MH086680-01A1 (NIH)
Record Dates: First submitted 2014-05-20; First posted 2014-05-22 (Estimated); Last update posted 2014-05-22 (Estimated); Status verified 2014-05

CONDITIONS: Depression
Keywords: Antepartum depressive symptoms; Antepartum depression; Cognitive behavioral intervention; Feasibility; randomized clinical trial
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Insight-Plus Cognitive Behavioral Intervention (Experimental): Insight-Plus is a 6-session, manualized, cognitive behavioral intervention (CBI) culturally tailored for a diverse group of rural low-income women at low and high risk for antepartum depression.
  Interventions: Behavioral: Insight-Plus Cognitive Behavioral Intervention
- Treatment as Usual (TAU) (No Intervention): Treatment as Usual (TAU) Control

INTERVENTIONS:
Behavioral: Insight-Plus Cognitive Behavioral Intervention — Insight-Plus is a 6-session, manualized, cognitive behavioral intervention (CBI) culturally tailored for a diverse group of rural low-income women at low and high risk for antepartum depression.
  Arms: Insight-Plus Cognitive Behavioral Intervention

SUMMARY:
The hypotheses were as follows:

H1. Women at low-moderate risk for APD at T1 (baseline EPDS scores of 5-9) in the cognitive behavioral intervention (CBI) group will maintain low-moderate risk status and have significantly fewer APD symptoms at T2 and T3 than women at low-moderate risk for APD in the (TAU) control group (as measured by percent of participants with EPDS scores <9 at T2 and T3 and mean score changes).

H2: Women at high risk for APD at T1 (baseline EPDS scores ≥10) in the CBI group will have a significantly greater reduction in APD symptoms at T2 and T3 than women at high risk for APD in the TAU control group (as measured by percent of participants with EPDS scores <10 at T2 and T3 and mean score changes).

DETAILED DESCRIPTION:
We collected data using Netbooks computers pre-programmed with Qualtrics survey forms.

At baseline (T1), post intervention (T2) and 1-month follow-up (T3), participants were administered the EPDS and the BDI-II and the Dolphin MINI neuropsychiatric Interview version 6. A similar time frame was used for the TAU group. Paired T-tests were used to determine mean change in EPDS scores (primary analysis) and BDI-II scores (secondary analysis) within each of the CBI and TAU groups at T2 and T3. A T-test measured differences in EPDS and BDI-II scores for the same time periods.

* The sample size was based on the PI's pilot intervention study. Using a conservative estimate of 500 eligible women from both sites per year at a 42% depression risk rate (moderate and high), and a 46% enrollment rate, it will be possible to accrue 97 subjects per year at risk for APD (moderate and high risk) or 193 subjects over the first 24 months of the study. Using the recruitment, retention, and eligibility patterns from the previous study, a total study sample of 124 subjects, 62 in the IP-CBI group and 62 in the TAU control group, allows for a 20% (24) drop-out rate and achieve the goal of 50 women in the IP-CBI and 50 women in the TAU control group.
* We planned to determine if there were significant differences in EPDS baseline scores in the CBI and TAU groups for the full sample and for the CBI and TAU groups stratified by high or low-moderate risk for antepartum depression.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Between 6-30 weeks pregnant
* Enrolled as a patient at the local health department (LHD) or Brody School of Medicine Regional Perinatal Center (BSOM-RPC)
* Self-identified as African American, Caucasian, or Hispanic
* Able to read at a 4th grade level;
* Have a or score >4 on the Edinburgh Postnatal Depression Scale (EPDS)
* Are willing to complete the informed consent form
* Enrolled in Medicaid or are low-income based on Women's Infant and Children (WIC) eligibility criteria.

Exclusion Criteria:

* Have had a spontaneous abortion before 20 weeks of pregnancy
* Diagnosed with schizophrenia or bipolar disorder with or without psychosis, or are currently receiving treatment for depression; or have an organic mental disorder
* Diagnosed with a high-risk pregnancy that requires bed rest or hospitalization-- Demonstrated an active suicidal plan
* Had a concurrent medical condition, such as hypothyroidism, that would explain depression.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2010-12; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Mean change in Edinburgh Postpartum Depression Scale (EPDS) Scores from baseline to post intervention and 1-month follow-up | Post-treatment and 1-month follow-up and an equivalent time frame for the TAU group
  Outcomes were mean change in Edinburgh Postpartum Depression Scale (EPDS) Scores in the CBI and TAU women from baseline (T1) to post-treatment (T2) and 1-month follow-up (T3) in those at low-moderate and high-risk for antepartum depression.

SECONDARY OUTCOMES:
Mean change in antepartum Beck Depression Inventory (BDI-II) Scores from baseline to post intervention and 1-month follow-up | Post-treatment and 1-month follow-up and an equivalent time frame for the TAU Group
  Outcomes were mean change in Beck Depression Inventory (BDI-II) Scores in the CBI and TAU women from baseline (T1) to post-treatment (T2) and 1-month follow-up (T3) in those at low-moderate and high-risk for antepartum depression.

OTHER OUTCOMES:
Mean change scores of mediators and moderators related to the EPDS | Post-treatment and 1-month follow-up and an equivalent time frame for the TAU group
  Mean change scores of mediators and moderators related to the EPDS mean T1-T2 and T1-T3 change scores within the CBI and the TAU control group

CONTACTS AND LOCATIONS:
Overall Officials: Darlene E Jesse, PhD, CNM, Principal Investigator — East Carolina University
Locations (2):
- United States (2):
  - Brody School of Medicine Regional Perinatal Center, Greenville, North Carolina
  - Pitt County Health Department, Greenville, North Carolina

REFERENCES:
- [Derived] Jesse DE, Gaynes BN, Feldhousen EB, Newton ER, Bunch S, Hollon SD. Performance of a Culturally Tailored Cognitive-Behavioral Intervention Integrated in a Public Health Setting to Reduce Risk of Antepartum Depression: A Randomized Controlled Trial. J Midwifery Womens Health. 2015 Sep-Oct;60(5):578-92. doi: 10.1111/jmwh.12308. Epub 2015 Aug 10. PMID 26261095